CLINICAL TRIAL: NCT00331812
Title: Study of Mitochondrial Functions and Oxidative Stress in ALS Patients.
Brief Title: Mitochondrial Functions and Oxidative Stress in ALS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Limoges (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Dr Corinne BOUTELOUP, CHU Clermont-Ferrand
Other Study IDs: CHU63-0007
Record Dates: First submitted 2006-05-23; First posted 2006-05-31 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Hypermetabolism; Mitochondrial abnormalities; Oxidant/antioxidant status
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Oxidative Stress

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Mitochondrial functions and oxidative stress

SUMMARY:
In Amyotrophic Lateral Sclerosis (ALS), malnutrition is frequent (16 to 50 % of the patients) and is an independent prognostic factor. One of the implicated factors is the increase of resting energy expenditure (REE) which can be found in about 50 % of ALS patients. The origin of this hypermetabolism is currently unknown but could be located in the mitochondria. In fact, some studies have found mitochondrial abnormalities and the existence of an oxidative stress. Thus, the aim of this study is to characterize the mitochondrial abnormalities and the oxidant/antioxidant status of ALS patients and to determine their relationship with the metabolic status, hypermetabolism or normometabolism. Three groups of patients will be studied : 20 hypermetabolic ALS patients, 20 normometabolic ALS patients and 20 healthy volunteers paired for age and sex.

DETAILED DESCRIPTION:
In Amyotrophic Lateral Sclerosis (ALS), malnutrition is frequent (16 to 50 % of the patients) and is an independent prognostic factor. One of the implicated factors is the increase of resting energy expenditure (REE) which can be found in about 50 % of ALS patients. The origin of this hypermetabolism is currently unknown but could be located in the mitochondria. In fact, some studies have found mitochondrial abnormalities and the existence of an oxidative stress. Thus, the aim of this study is to characterize the mitochondrial abnormalities and the oxidant/antioxidant status of ALS patients and to determine their relationship with the metabolic status, hypermetabolism or normometabolism. Three groups of patients will be studied : 20 hypermetabolic ALS patients, 20 normometabolic ALS patients and 20 healthy volunteers paired for age and sex.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age > 30 years
* definite or probable ALS according to the El Escorial criteria, bulbar or spinal form, ALS diagnosis < 1 year and treatment by riluzole.

Exclusion Criteria:

* family history of ALS,
* oral, enteral or parenteral nutritional supply,
* vitamin or trace element supplementation
* confusing illness (cancer, diabetes, chronic infectious or inflammatory disease,thyroid disorders, recent surgery...),
* current tobacco use,
* alcoholism
* treatment by corticosteroids,
* diuretics,
* anorectics
* NSAIDs
* cytotoxics
* anticoagulants...

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of patients will be studied : 20 hypermetabolic ALS patients, 20 normometabolic ALS patients and 20 healthy volunteers paired for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-02; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
relationship between these abnormalities and the metabolic status (hypermetabolism or normometabolism).

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Bouteloup, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Desport JC, Preux PM, Magy L, Boirie Y, Vallat JM, Beaufrere B, Couratier P. Factors correlated with hypermetabolism in patients with amyotrophic lateral sclerosis. Am J Clin Nutr. 2001 Sep;74(3):328-34. doi: 10.1093/ajcn/74.3.328. PMID 11522556
- [Background] Ferrante RJ, Browne SE, Shinobu LA, Bowling AC, Baik MJ, MacGarvey U, Kowall NW, Brown RH Jr, Beal MF. Evidence of increased oxidative damage in both sporadic and familial amyotrophic lateral sclerosis. J Neurochem. 1997 Nov;69(5):2064-74. doi: 10.1046/j.1471-4159.1997.69052064.x. PMID 9349552
- [Background] Menzies FM, Ince PG, Shaw PJ. Mitochondrial involvement in amyotrophic lateral sclerosis. Neurochem Int. 2002 May;40(6):543-51. doi: 10.1016/s0197-0186(01)00125-5. PMID 11850111